CLINICAL TRIAL: NCT00934323
Title: An Open, Randomized, Two-Treatment, Crossover Study to Assess the Dose Proportionality of Glimepiride Between Amaryl M SR 1/500mg and 2/500mg (Glimepiride-Metformin Fixed Dose Combination Tablet) in Healthy Male Subjects
Brief Title: Dose Proportionality Study About Amaryl M Slow Release (SR) 1/500 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Hye Jin Cheong/ Head of Clinical Research Operation, Handok Pharmaceuticals, Co., Ltd
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: M_SR_001
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
Keywords: volunteer
MeSH Terms: interventions — glimepiride; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TR sequential group (Experimental): Amaryl M SR 1/500 mg in period 1 and Amaryl M SR 2/500 mg in period 2
  Interventions: Drug: Amaryl M SR 1/500 mg; Drug: Amaryl M SR 2/500 mg
- RT sequential group (Active Comparator): Amaryl M SR 2/500 mg in period 1 and Amaryl M SR 1/500 mg in period 2
  Interventions: Drug: Amaryl M SR 1/500 mg; Drug: Amaryl M SR 2/500 mg

INTERVENTIONS:
Drug: Amaryl M SR 1/500 mg — single oral administration in period 1 for TR sequential group, and in period 2 for RT sequential group
  Other Names: Amaryl Mex 1/500mg, glimepiride 1mg & metformin HCl 500mg
Drug: Amaryl M SR 2/500 mg — single oral administration in period 2 for TR sequential group, and in period 2 for RT sequential group
  Other Names: Amaryl Mex 2/500mg, glimepiride 2mg & metformin HCl 500mg

SUMMARY:
The pharmacokinetics of glimepiride and metformin will be compared after single dose intake of both combinations in order to answer to the following questions:

* Is there a dose proportionality effect between Amaryl M SR 1/500 mg and Amaryl M SR 2/500 mg?
* What is the safety profile of Amaryl M SR 1/500 mg and Amaryl M SR 2/500 mg?

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 20 to 45 years of age, inclusive (Age based on the date to give the informed consent)
* Ideal body weight (Broca index): between 50 to 90 kg, inclusive, and within ±20 % of Ideal Body Weight, [(Height in cm-100)×0.9]
* Subjects who are appropriate to participate in this study judged from clinical laboratory and physical examinations taken within 4weeks prior to the start of study
* Subjects who are able to abstain from caffein or caffein-containing products (e.g., coffee, cola, tea, chocolate), grapefruit and grapefruit containing products, alcohol and smoking within 72 hours before dosing and during the hospitalization
* Subjects who are reliable and willing to make themselves available during the study period, are willing to follow the study protocol, and give their written informed consent voluntarily

Exclusion Criteria:

* History of allergies including drug allergy, except untreated, asymptomatic, seasonal allergies at the time of dosing
* Use any prescriptive medication, Korean traditional medication not considered acceptable by the clinical investigator during the last 10 days period before first dosing, or use any OTC medication not considered acceptable by the clinical investigator during the last 7 days period before first dosing (If used medication is considered acceptable by investigator, patients can be included)
* History of significant clinical illness needs medical caution, including cardiovascular, immunologic, hematologic, neuropsychiatric, respiratory, gastrointestinal, hepatic, or renal disease or other chronic disease
* History of a significant surgical resection of gastrointestinal tract except appendectomy
* Abnormal clinical laboratory findings, especially for AST or ALT> 1.25 fold of upper normal limit
* Evidence of alcohol abuse (defined as regular alcohol intake that exceeds 24 oz [675 ml] of beer, 12 oz [340 ml] of wine or 160 ml of soju or 3 oz [85 ml] hard liquor [e.g., brandy, whiskey, gin] per day) or drug abuse
* Heavy smokers (> 10 cigarettes per day), or can't quit smoking during hospitalization
* Participation in clinical trials of any drug within 3 months prior to the participation of the study
* Donation of whole blood within 2 months or a unit of blood within 1 month prior to the start of study [Day 1].
* Positive Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCV Ab), or HIV antibody
* Judged to be inappropriate for the study by the investigator

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
AUClast/D, Cmax/D | pre-dose (=1d 0h), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24 hrs after drug administration

SECONDARY OUTCOMES:
Tmax, T1/2 | pre-dose (=1d 0h), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24 hrs after drug administration
Vital signs, ECG, physical examination, clinical laboratory tests | screening, treatment period 1 & 2, Post-study visit
Adverse Event | Treatment period 1 & 2, Post-study visit

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, Professor, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Shin KH, Kim SE, Yoon SH, Cho JY, Jang IJ, Shin SG, Yu KS. Pharmacokinetic comparison of a new sustained-release formulation of glimepiride/metformin 1/500 mg combination tablet and a sustained-release formulation of glimepiride/metformin 2/500 mg combination tablet in healthy Korean male volunteers: a randomized, 2-sequence, 2-period, 2-treatment crossover study. Clin Ther. 2011 Nov;33(11):1809-18. doi: 10.1016/j.clinthera.2011.10.003. Epub 2011 Oct 27. PMID 22036245